CLINICAL TRIAL: NCT03165526
Title: The AMPLATZER™ Post-infarct Muscular VSD Occluder Humanitarian Device Exemption (H070005) Post Approval Study
Acronym: PIVSD PAS
Status: Completed | Type: Observational
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Other Study IDs: SJM-CIP-10191
Record Dates: First submitted 2017-05-06; First posted 2017-05-24 (Actual); Results first posted 2024-10-10 (Actual); Last update posted 2024-10-10 (Actual); Status verified 2024-07

CONDITIONS: Post-Infarction Ventricular Septal Defect

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (2):
- First Cohort: All available Emergency and Compassionate PIVSD Occluder subject data from 2011 until the end of 2016 will be utilized to determine technical success and acute survival. All subjects belonging to this cohort must have undergone an attempt to close a post-infarct VSD using the AMPLATZER™ PIVSD Occluder.
  Interventions: Device: AMPLATZER™ Post-infarct Muscular VSD Occluder
- Second Cohort: This cohort will consist of subjects over the age of 18 years who have previously been successfully implanted with the PIVSD Occluder and
  * For living subjects, the subject or subject's legally authorized representative has provided consent to participate in this study.
  * Subject's post-procedure echocardiogram is evaluable and can be sent to the echocardiography core laboratory for residual shunt assessment.
  Therefore, this cohort will be composed of retrospectively enrolled subjects. This cohort will be utilized to determine acute and chronic closure and chronic survival.
  Interventions: Device: AMPLATZER™ Post-infarct Muscular VSD Occluder

INTERVENTIONS:
Device: AMPLATZER™ Post-infarct Muscular VSD Occluder — The AMPLATZER™ PIVSD Occluder is intended for percutaneous transcatheter closure of post-myocardial infarct muscular VSDs in patients who are not satisfactory surgical candidates.

SUMMARY:
FDA issued a Humanitarian Device Exemption (HDE) approval order for the AMPLATZER™ PIVSD Occluder (H070005) on January 10, 2017. The Conditions of Approval require that SJM conduct a post approval study to evaluate the safety and probable benefit of the AMPLATZER™ PIVSD Occluder.

DETAILED DESCRIPTION:
This is a multi-center, observational study to evaluate the safety and probable benefit of the AMPLATZER™ PIVSD Occluder for use in transcatheter closure of muscular ventricular septal defects following a myocardial infarction in the post approval setting.

The study has five endpoints (safety: acute and chronic survival; effectiveness: technical success, acute and chronic closure).Two cohorts will be utilized to obtain study endpoint data. The first cohort will be comprised of all available Emergency and Compassionate PIVSD Occluder subject data from 2011 until the end of 2016 and these data will be used to determine technical success and acute survival. The second cohort of thirty subjects will be comprised of patients who are successfully implanted with a PIVSD Occluder from 2011 onward at activated study centers. The index procedure must have occurred >6 months prior to enrollment. Subject identification will occur until data on a minimum of 30 subjects with PIVSD Occluders for post myocardial infarct VSD and post-procedure echocardiogram available for evaluation of residual shunt by the echocardiography core laboratory have been enrolled. The thirty subject cohort data will be used to determine acute closure, chronic closure, and chronic survival endpoints.

The study will be conducted at up to 50 centers in the U.S. The expected duration of enrollment is approximately 4 years. The total duration of the clinical study is expected to be 4.5 years.

ELIGIBILITY:
First Cohort:

Patients who have undergone an attempt to close a post-infarct VSD using the AMPLATZER™ PIVSD Occluder via Emergency and Compassionate 2011 until the end of 2016.

Second Cohort:

* Over 18 years old
* Patients who have previously been successfully implanted with the AMPLATZER™ PIVSD Occluder
* For living subjects, the subject or subject's legally authorized representative has provided consent to participate in this study
* Subject's post-procedure echocardiogram is evaluable and can be sent to the echocardiography core laboratory for residual shunt assessment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: First Cohort: Patients who have undergone an attempt to close a post-infarct VSD using the AMPLATZER™ PIVSD Occluder via Emergency and Compassionate 2011 until the end of 2016.
  Second Cohort: This cohort will consist of subjects over the age of 18 years who have previously been successfully implanted with the AMPLATZER™ PIVSD Occluder.
Sampling Method: Non-Probability Sample
Enrollment: 131 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2021-11-29 (Actual); Study Completion 2021-11-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ryan Palmer, Study Director — Sponsor GmbH
Locations (17):
- United States (17):
  - University of California at San Francisco, San Francisco, California
  - Shands at the University of Florida, Gainesville, Florida
  - Johns Hopkins University Hospital, Baltimore, Maryland
  - Spectrum Health Butterworth Hospital, Grand Rapids, Michigan
  - University of Minnesota Medical Center Fairview, Minneapolis, Minnesota
  - Buffalo General Hospital, Buffalo, New York
  - Lenox Hill Hospital, New York, New York
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Duke University, Durham, North Carolina
  - UNC Regional Physicians Carolina Cardiology, High Point, North Carolina
  - Good Samaritan Trihealth Hospital, Cincinnati, Ohio
  - Memorial Hermann Hospital, Houston, Texas
  - Baylor Scott & White, Plano, Texas
  - Swedish Medical Center, Seattle, Washington
  - Providence Medical Research Group, Spokane, Washington
  - University of Wisconsin Hospital and Clinics, Madison, Wisconsin
  - Marshfield Clinic, Marshfield, Wisconsin

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Second Cohort: This cohort will consist of subjects over the age of 18 years who have previously been successfully implanted with the PIVSD Occluder and
  * For living subjects, the subject or subject's legally authorized representative has provided consent to participate in this study.
  * Subject's post-procedure echocardiogram is evaluable and can be sent to the echocardiography core laboratory for residual shunt assessment.
  Therefore, this cohort will be composed of retrospectively enrolled subjects. This cohort will be utilized to determine acute and chronic closure and chronic survival.
  AMPLATZER™ Post-infarct Muscular VSD Occluder: The AMPLATZER™ PIVSD Occluder is intended for percutaneous transcatheter closure of post-myocardial infarct muscular VSDs in patients who are not satisfactory surgical candidates.
Period: Overall Study
Arm/Group | First Cohort | Second Cohort
Started | 99 | 32
Completed | 99 | 32
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Amplatzer Post-Infarct Muscular VSCD Occluder Humanitarian Device Exemption Post-Approval Study: Cohort 1: All available Emergency and Compassionate PIVSD Occluder subject data from 2011 until the end of 2016 will be utilized to determine technical success and acute survival. All subjects belonging to this cohort must have undergone an attempt to close a post-infarct VSD using the AMPLATZER™ PIVSD Occluder.
  Cohort 2: This cohort will consist of subjects over the age of 18 years who have previously been successfully implanted with the PIVSD Occluder and
  * For living subjects, the subject or subject's legally authorized representative has provided consent to participate in this study.
  * Subject's post-procedure echocardiogram is evaluable and can be sent to the echocardiography core laboratory for residual shunt assessment.
  Therefore, this cohort will be composed of retrospectively enrolled subjects. This cohort will be utilized to determine acute and chronic closure and chronic survival.
  AMPLATZER™ Post-infarct Muscular VSD Occluder: The AMPLATZER™ PIVSD Occluder is intended for percutaneous transcatheter closure of post-myocardial infarct muscular VSDs in patients who are not satisfactory surgical candidates.
Arm/Group | Amplatzer Post-Infarct Muscular VSCD Occluder Humanitarian Device Exemption Post-Approval Study
Number analyzed (Participants) | 131
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: The PIVSD post-approval study composed of 2 cohorts including Cohort 1 (n=99) and Cohort 2 (n=32).
  years
    Cohort 1: number analyzed (Participants) | 99
    Cohort 1 | 68.6 (11.9)
    Cohort 2: number analyzed (Participants) | 32
    Cohort 2 | 66.4 (10.9)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: The PIVSD post-approval study composed of 2 cohorts including Cohort 1 (n=99) and Cohort 2 (n=32)
  Participants
    Cohort 1: number analyzed (Participants) | 99
    Cohort 1: Female | 46
    Cohort 1: Male | 53
    Cohort 2: number analyzed (Participants) | 32
    Cohort 2: Female | 15
    Cohort 2: Male | 17
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: The PIVSD post-approval study composed of 2 cohorts including Cohort 1 (n=99) and Cohort 2 (n=32). Ethnicity was not collected for Cohort 1.
  Participants
    Cohort 1: number analyzed (Participants) | 0
    Cohort 2: number analyzed (Participants) | 32
    Cohort 2: Hispanic or Latino | 2
    Cohort 2: Not Hispanic or Latino | 25
    Cohort 2: Unknown or Not Reported | 5
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: The PIVSD post-approval study composed of 2 cohorts including Cohort 1 (n=99) and Cohort 2 (n=32). Race was not collected for Cohort 1.
  Participants
    Cohort 1: number analyzed (Participants) | 0
    Cohort 2: number analyzed (Participants) | 32
    Cohort 2: American Indian or Alaska Native | 0
    Cohort 2: Asian | 0
    Cohort 2: Native Hawaiian or Other Pacific Islander | 0
    Cohort 2: Black or African American | 1
    Cohort 2: White | 27
    Cohort 2: More than one race | 0
    Cohort 2: Unknown or Not Reported | 4
Region of Enrollment [Count of Participants; unit: Participants]
  United States: Cohort 1 | 99
  United States: Cohort 2 | 32
Location of MI [Count of Participants; unit: Participants] — Population: The PIVSD post-approval study composed of 2 cohorts including Cohort 1 (n=99) and Cohort 2 (n=32).
  Participants
    Cohort 1: number analyzed (Participants) | 99
    Cohort 1: Anterior (LAD) | 39
    Cohort 1: Posterior/Inferior (RCA) | 47
    Cohort 1: Lateral (Cicumflex) | 2
    Cohort 1: Unknown | 11
    Cohort 2: number analyzed (Participants) | 32
    Cohort 2: Anterior (LAD) | 14
    Cohort 2: Posterior/Inferior (RCA) | 16
    Cohort 2: Lateral (Cicumflex) | 1
    Cohort 2: Unknown | 1
Weight (kg) [Mean (Standard Deviation); unit: kg] — Population: The PIVSD post-approval study composed of 2 cohorts including Cohort 1 (n=99) and Cohort 2 (n=32). Weight was not collected for Cohort 1.
  kg
    Cohort 1: number analyzed (Participants) | 0
    Cohort 2: number analyzed (Participants) | 32
    Cohort 2 | 81.48 (16.76)
Height (cm) [Mean (Standard Deviation); unit: cm] — Population: The PIVSD post-approval study composed of 2 cohorts including Cohort 1 (n=99) and Cohort 2 (n=32).
  cm
    Cohort 1: number analyzed (Participants) | 0
    Cohort 2: number analyzed (Participants) | 31
    Cohort 2 | 168.47 (9.30)
BMI [Mean (Standard Deviation); unit: kg/m^2] — Population: The PIVSD post-approval study composed of 2 cohorts including Cohort 1 (n=99) and Cohort 2 (n=32). BMI was not collected for Cohort 1. Data was available for 31/32 of Cohort 2 subjects.
  kg/m^2
    Cohort 1: number analyzed (Participants) | 0
    Cohort 2: number analyzed (Participants) | 31
    Cohort 2 | 28.34 (5.62)
Medical History [Count of Participants; unit: Participants] — Population: The PIVSD post-approval study composed of 2 cohorts including Cohort 1 (n=99) and Cohort 2 (n=32). Medical History was not collected for Cohort 1. Data was available for 29 and 31 of the Cohort 2 subjects for hyperlipidemia and history of smoking, respectively.
  Participants
    Cohort 1: number analyzed (Participants) | 0
    Cohort 2 - Hypertension: number analyzed (Participants) | 32
    Cohort 2 - Hypertension | 21
    Cohort 2 - Diabetes: number analyzed (Participants) | 32
    Cohort 2 - Diabetes | 10
    Cohort 2 - Hyperlipidemia: number analyzed (Participants) | 29
    Cohort 2 - Hyperlipidemia | 19
    Cohort 2 - History of Smoking: number analyzed (Participants) | 31
    Cohort 2 - History of Smoking | 18

OUTCOME MEASURES:

1. Primary Outcome: Effectiveness Endpoint 1: Technical Success
Description: Technical success occurs when a subject is successfully implanted with a PIVSD device in the ventricular septal defect. An implant attempt occurs when the delivery system is inserted in the subject's vasculature.
Time Frame: End of Implant Procedure
Population: The analysis population includes all Emergency and Compassionate PIVSD subjects who have an attempted device placement (defined as the delivery system enters the subject's vasculature in an attempt to place a device) from 2011 until the end of 2016.
Measure: Count of Participants; unit: Participants
Groups:
- Cohort 1: Cohort 1 consisted of all Emergency and Compassionate PIVSD subjects who have an attempted device placement (defined as the delivery system enters the subject's vasculature in an attempt to place a device) from 2011 until the end of 2016 (n=99).
Arm/Group | Cohort 1
Number analyzed (Participants) | 99
Participants | 76

2. Primary Outcome: Effectiveness Endpoint 2: Acute Closure
Description: Acute closure is defined as the absence of a residual shunt ≥3 mm, and will be assessed based on an echocardiogram obtained immediately after the successful deployment of the device and up to 7 days post-procedure.
Time Frame: Up to 7 days post-procedure
Population: The analysis population will include all enrolled subjects, i.e., this population will include subjects from Cohort 2 which will be comprised of subjects who have previously been successfully implanted with the PIVSD Occluder, the subject's post-procedure echocardiogram is able to be evaluated for residual shunt by the echocardiography core laboratory, and, for living subjects, informed consent has been obtained.
Measure: Count of Participants; unit: Participants
Groups:
- Cohort 2: Cohort 2: This cohort will consist of subjects over the age of 18 years who have previously been successfully implanted with the PIVSD Occluder and
  * For living subjects, the subject or subject's legally authorized representative has provided consent to participate in this study.
  * Subject's post-procedure echocardiogram is evaluable and can be sent to the echocardiography core laboratory for residual shunt assessment.
Arm/Group | Cohort 2
Number analyzed (Participants) | 32
Participants | 17

3. Primary Outcome: Effectiveness Endpoint 3: Chronic Closure
Description: Chronic closure is defined as the absence of a residual shunt ≥3 mm at 6 months or later.
Time Frame: 6 months or later following a PIVSD device implant through study completion, an average of 1 year
Population: The analysis population will include enrolled subjects from Cohort 2 with an implanted PIVSD device who have a 6-months or later post-procedure echocardiogram available for review.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 2
Number analyzed (Participants) | 6
Participants | 4

4. Primary Outcome: Safety Endpoint 1: Acute Survival
Description: Acute survival is defined as survival for at least 24 hours following an attempted PIVSD device implant.
Time Frame: Equal to or greater than 24 hours following an attempted PIVSD device implant through study completion, up to 9.7 years post-procedure
Population: The analysis population will include all Emergency and Compassionate PIVSD subjects who have an attempted device placement from 2011 until the end of 2016 but will exclude subjects whose survival status is not known through at least 24 hours after the procedure.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1
Number analyzed (Participants) | 89
Participants | 75

5. Primary Outcome: Safety Endpoint 2: Chronic Survival
Description: Chronic survival is defined as survival for at least 183 days from the time of first successful implant.
Time Frame: Equal to or greater than 183 days from the time of first successful implant through study completion, up to 9.7 years post-procedure
Population: The analysis will be conducted on both cohorts. The first analysis population is Cohort 1(all Emergency and Compassionate PIVSD subjects who have an attempted device placement from 2011 until the end of 2016). The second analysis population is Cohort 2 (those previously implanted with the PIVSD Occluder, provided informed consent (for living subjects only), and the subject's post-procedure echocardiogram is able to be evaluated for residual shunt by the echocardiography core laboratory).
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Cohort 2: Cohort 2 consists of subjects who have been previously implanted with the PIVSD Occluder
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 99 | 32
percentage of participants | 37.2 [27.0 to 47.3] | 46.4 [27.9 to 63.1]

ADVERSE EVENTS:
Time Frame: Data in this study were collected retrospectively; therefore, no adverse event information was collected. Additionally, these data do not apply towards any of the study endpoints. Mortality data was collected to estimate survival through study completion, up to 9.7 years post-procedure.
Description: Data in this study were collected retrospectively; therefore, no adverse event information was collected. Additionally, these data do not apply towards any of the study endpoints. Mortality data was collected to estimate survival through study completion, up to 9.7 years post-procedure.
Groups:
- Cohort 1: Cohort 1: All available Emergency and Compassionate PIVSD Occluder subject data from 2011 until the end of 2016 will be utilized to determine technical success and acute survival. All subjects belonging to this cohort must have undergone an attempt to close a post-infarct VSD using the AMPLATZER™ PIVSD Occluder.
- Cohort 2: Cohort 2: This cohort will consist of subjects over the age of 18 years who have previously been successfully implanted with the PIVSD Occluder and
  * For living subjects, the subject or subject's legally authorized representative has provided consent to participate in this study.
  * Subject's post-procedure echocardiogram is evaluable and can be sent to the echocardiography core laboratory for residual shunt assessment.
  Therefore, this cohort will be composed of retrospectively enrolled subjects. This cohort will be utilized to determine acute and chronic closure and chronic survival.
Arm/Group | Cohort 1 | Cohort 2
All-Cause Mortality (participants affected / at risk) | 59/99 | 16/32
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-12-11): https://cdn.clinicaltrials.gov/large-docs/26/NCT03165526/Prot_SAP_000.pdf